CLINICAL TRIAL: NCT07018752
Title: A Platform Trial, Evaluating New Drugs or Combination in Relapsed or Refractory Peripheral T-cell Lymphomas
Brief Title: A Platform Trial Evaluating New Drugs or Combination in R/R Peripheral T-cell Lymphomas
Acronym: PlaTform
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: iOnctura (Industry); AbbVie (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PlaTform; 2024-514954-63 (EudraCT Number)
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-06

CONDITIONS: Peripheral T Cells Lymphoma (PTCL)
Keywords: lymphoma; peripheral T cells lymphoma; roginolisib; azacitidine; refractory peripheral T-cells lymphoma; relapsed peripheral T-cells lymphoma; golcadomide
MeSH Terms: conditions — Lymphoma | interventions — Azacitidine

STUDY DESIGN:
Intervention Model Description: Multiples arms/sub-studies will be opened in parallel and/or successively. The number of arms/sub-studies will be increasing throughout the study and is not a fixed number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Origina-ly-T (Experimental): Open-label phase 2 sub-study to evaluate the efficacy and safety of roginolisib in relapsed/refractory peripheral T-cells lymphoma. Study treatment will be administered until unacceptable toxicity, disease progression, subject/physician decision to withdraw, whichever happens first.
  31 evaluable patients needed.
  Interventions: Drug: roginolisib
- GolcAza (Experimental): Open-label phase 1 sub-study to identify the maximum tolerated dose of golcadomide in association with oral 5-azacitidine and evaluate the efficacy and safety of the determined combination of oral 5-azacitidine and golcadomide in relapsed/refractory follicular helper T-cell lymphoma subjects.
  Subjects will receive golcadomide and oral 5-azacitidine until end of study or until disease progression, unacceptable toxicity, subject/physician decision to withdraw, whichever occurs first.
  Minimum 18 evaluable patient required.
  Interventions: Drug: golcadomide; Drug: azacitidine

INTERVENTIONS:
Drug: roginolisib — Roginolisib daily intake
  Arms: Origina-ly-T
Drug: golcadomide — Golcadomide daily intake
  Arms: GolcAza
Drug: azacitidine — oral 5-azacitidine daily intake
  Arms: GolcAza

SUMMARY:
This study is a platform trial for the evaluation of new drugs or combination of drugs in relapsed or refractory peripheral T-cell lymphomas.

The objective of the study is to generate exploratory data on new drugs or combination of drugs to treat refractory/relapse peripheral T-cells lymphoma to better identify the population of interest and design future correct clinical trials.

Primary objectives of the different sub-studies :

* phase 1 sub-studies: determine the safety and tolerability of escalating doses of the sub-study treatment
* phase 2 sub-studies: identify drugs that will improve significantly the outcome in target patients Secondary objectives of both sub-studies: analyze the response rate, the clinical benefit rate, the progression-free survival, the duration of response, the time to next treatment or death, the overall survival, the rate of transplantation following study treatment and the safety profile of the drugs used

DETAILED DESCRIPTION:
This study is a platform trial evaluating new drugs or combination of drugs in relapsed or refractory peripheral T-cell lymphomas via multiple sub-studies. For phase 1 sub-studies, at least 18 evaluable patients are required per each sub-study. For phase 2 sub-studies, 31 evaluable patients are required per sub-study.

Each sub-study has its own specificities:

* Origina-ly-T: open-label phase 2 study evaluating the efficacy and safety of roginolisib in relapsed/refractory peripheral T-cells lymphoma. Study treatment will be administered until unacceptable toxicity, disease progression, subject/physician decision to withdraw, whichever happens first.
* GolcAza: open-label phase 1 study to identify the maximum tolerated dose of golcadomide in association with oral 5-azacitidine and evaluate the efficacy and safety of the determined combination of oral 5-azacitidine and golcadomide in relapsed/refractory follicular helper T-cell lymphoma subjects. Subjects will receive golcadomide and oral 5-azacitidine until end of study or until disease progression, unacceptable toxicity, subject/physician decision to withdraw, whichever occurs first.

ELIGIBILITY:
1. Subject who understood and voluntarily signed and dated an informed consent prior to any study-specific assessments/procedures being conducted;
2. Subject is ≥ 18 years of age at the time of signing the informed consent form (ICF);
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements;
4. Subject with histologically proven peripheral T-cell lymphoma according to the criteria of the WHO classification 2017 or 2022 (subjects with mycosis fungoides, Sezary syndrome, lymphoblastic or large granular lymphocytic lymphoma will be excluded). Tumor tissue (initial diagnosis or relapse) should be available for central pathology review and biological characterization;
5. Subject in relapse/refractory situation;
6. ECOG performance status 0 to 2, or 3 if thought to be related to lymphoma;
7. Adequate bone marrow function as defined by:

   * Absolute Neutrophil Count ≥ 1,5 x 10^9/L (≥ 1 x 10^9/L if related to lymphoma)
   * Platelets ≥ 75 x 10^9/L (≥ 50 x 10^9/L if related to lymphoma)
   * Hemoglobin ≥ 8 g/dL;
8. Anticipated life expectancy at least 3 months;
9. Presence of disease specific criteria allowing response evaluation. Unless otherwise specified, such criteria include:

   1. Baseline fluorodeoxyglucose PET-scan demonstrating at least one positive (FDG-avid) lesion;
   2. and at least one bi-dimensionally measurable nodal lesion, defined as > 1.5 cm in its longest dimension, or at least one bi-dimensionally measurable extra nodal lesion, defined as > 1.0 cm in its longest dimension;
10. Contraception:

    * For women of childbearing potential (WOCBP): must have a negative result for pregnancy test, at screening and within 24 hours prior to initiating study treatment. The WOCBP agree to abstain from becoming pregnant or breastfeeding, to remain abstinent (from heterosexual intercourse) or use at least one highly effective method of contraception and to refrain from donating eggs, during the treatment period (including periods of treatment interruption) and for at least the delay described in the sub-protocol for the concerned molecules;
    * For men of reproductive potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use at least a condom as method of contraception with a non-pregnant female partner of childbearing potential or a pregnant female partner, and to refrain from donating sperm, during the treatment period (including periods of treatment interruption), and for at least the delay described in the sub-protocol for the concerned molecules;
11. Subject covered by a social security system;
12. Subject who understands and speaks one of the country official languages unless local regulation authorizes independent translators;

    Additional inclusion criteria specific to Origina-ly-T sub-study:
13. For anaplastic large cell lymphoma subjects: failed or ineligible or intolerant to brentuximab vedotin. For extranodal NK/T-cells lymphoma: failed or ineligible or intolerant to asparaginase-containing regimen;

    Additional inclusion criteria specific to Golcaza sub-study:

13. Subject had local diagnosed (nodal) follicular helper T cell lymphoma according to WHO classification 2022 or ICC 2022 classification based on a surgical lymph node biopsy or needle core biopsy including any one of the following type:

* angioimmunoblastic type (AITL)
* follicular T cell type
* not otherwise specified (NOS);

  14. ECOG performance status 0 to 1 (supersedes criterium 6 of the Master protocol);

  15. Subjects must have an international normalized ratio (INR) < 1.5 x ULN and partial thromboplastin time (aPTT) < 1.5 x ULN (for subjects not receiving therapy). Note: Subjects receiving therapy for a thromboembolic event that occurred > 3months prior to enrollment are eligible as long as they are on a stable regimen of anticoagulation with warfarin, low-molecular weight heparin, or other approved therapeutic anticoagulation or antiplatelet regimen;

  16. Contraception (supersedes criterium 10 of the Master protocol):
* For women of childbearing potential (WOCBP): must have a negative result for pregnancy test, 10 to 14 days prior to initiating study treatment and within 24 hours prior to initiating study treatment. WOCBP agree to abstain from becoming pregnant or breastfeeding and to remain abstinent (refrain from heterosexual intercourse) or use two adequate methods of contraception, including at least one highly effective method of contraception , at least 28 days before the first dose of study treatment , during the treatment period (including periods of treatment interruption), and for at least 28 days after the last dose of golcadomide, and 6 months after the last dose of azacitidine. Women must refrain from donating eggs during this same period;
* For men: during the treatment period (including periods of treatment interruption), and for at least 28 days after the last dose of golcadomide and 3 months after the last dose of oral 5-azacitidine male subjects must:

  * With female partners of childbearing potential: use a condom associated with a highly effective method of contraception or remain abstinent (refrain from heterosexual intercourse)
  * With pregnant female partners: use a condom or remain abstinent (refrain from heterosexual intercourse) Men must refrain from donating sperm during this same period;

Exclusion Criteria:

1. Evidence of central nervous system involvement by lymphoma;
2. Any significant medical conditions, laboratory abnormality or psychiatric illness likely to interfere with participation in this clinical study (according to the investigator's decision);
3. Uncontrolled systemic fungal, bacterial, or viral infection;
4. Known Hepatitis C Virus (HCV) or active Hepatitis B Virus (HBV) infection defined as subject with detectable viral load (respectively detectable viral RNA or detectable viral DNA);
5. Active malignancy other than the one treated in this research, unless the subject has been free of the disease for 2 years (subjects with a history of a completely resected non-melanoma skin cancer or successfully treated for an in-situ carcinoma are eligible);
6. Use of any standard or experimental anti-cancer drug therapy within 28 days or a minimum of 5 half-lives of the drug, whatever the shortest prior to first administration of study drug;.
7. Subject taking corticosteroids within 14 days prior to first administration of study drug, unless administered at a cumulated dose equivalent of prednisone ≤ 20mg /day (within these 14 days);
8. Subject with prior autologous hematopoietic cell transplantation (auto-HCT) ≤ 3 months prior to starting investigational product(s). If subject had autologous SCT (Stem Cell Transplant) > 3 months prior to the start of investigational product(s), any unresolved (Grade > 1) autologous SCT-related toxicity;
9. Subject with prior allogeneic hematopoietic cell transplantation (allo-HCT) with either standard or reduced intensity conditioning ≤ 3 months prior to starting investigational product(s). If subject had allogeneic SCT > 3 months prior to the start of investigational product(s) and still has any unresolved situation including (Grade > 1) treatment-related toxicity and/or ongoing immunosuppressor therapy and/or more than mild (NIH consensus) chronic graft-versus-host disease;
10. Subject with major surgery ≤ 14 days prior to starting investigational product(s). Subjects must have recovered from any clinically significant effects of recent surgery;
11. Subject who has received prior localized anticancer therapy (eg. radiotherapy [including palliative radiotherapy]) ≤ 14 days prior to starting investigational product(s);
12. Known or suspected hypersensitivity to active substance or to any of the excipients;
13. Pregnant, planning to become pregnant, or lactating woman;
14. Person deprived of his/her liberty by a judicial or administrative decision;

    Exclusion criteria specific to Origina-ly-T sub-study:
15. Positive HIV test at screening, with the following exception: individuals with a positive HIV test at screening are eligible provided they are stable on antiretroviral therapy for at least 4 weeks, have a CD4 count ≥ 200/uL, have an undetectable viral load, and have not had a history of opportunistic infection attributable to HIV within the last 12 months
16. Impaired renal function (calculated CKP-EPI, MDRD or Cockcroft-Gault Creatinine Clearance < 30 ml/min) or impaired liver function tests (serum total bilirubin level > 34 μmol/L), except in case of Gilbert's Syndrome, or documented liver or pancreatic involvement by lymphoma, serum transaminases (AST or ALT) > 3 upper normal limits, unless elevated to up to 5 x ULN due to peripheral T-cells lymphoma);
17. Significant cardiovascular disease [e.g., Objective Class C or D heart diseases (cf. Classes of Heart Failure | American Heart Association)], myocardial infarction within the previous 6 months, unstable arrhythmia, or unstable angina);
18. Prior exposure to PI3Kdelta inhibitor;
19. Known or suspected allergies, hypersensitivity, or intolerance to Roginolisib or its excipients;
20. Inability to swallow food or any condition of the upper gastrointestinal tract that precludes administration of oral medications;
21. Subjects with a diagnosis of cutaneous T-cell lymphoma (CTCL);
22. Prior solid organ transplantation;

Exclusion criteria specific to GolcAza sub-study:

15. Evidence of positive HTLV1 serology;

16. Positive HIV test at screening, with the following exception: individuals with a positive HIV test at screening are eligible provided they are stable on antiretroviral therapy for at least 4 weeks, have a CD4 count ≥ 200/uL, have an undetectable viral load, and have not had a history of opportunistic infection attributable to HIV within the last 12 months;

17. Impaired renal function (calculated CKD-EPI, MDRD or Cockcroft-Gault Creatinine Clearance < 30 ml/min) or impaired liver function tests (serum total bilirubin level > 34 μmol/L) except in case of Gilbert's Syndrome, or documented liver or pancreatic involvement by lymphoma, serum transaminases (AST or ALT) > 3 upper normal limits (except documented liver involvement by lymphoma);

18. Prior exposure to golcadomide;

19. Refractory to azacitidine;

20. Significant cardiovascular disease [e.g., Objective Class C or D heart diseases (cf. Classes of Heart Failure | American Heart Association)], myocardial infarction ≤ 3 months prior to starting golcadomide, unstable angina pectoris ≤ 3 months prior to starting golcadomide), or complete left bundle branch or bifascicular block), congenital long QT syndrome, QTcF ≥ 470 msec on screening, persistent or clinically meaningful ventricular arrhythmias;

21. Received strong CYP3A inhibitors, moderate CYP3A inhibitors, strong CYP3A inducers, moderate CYP3A inducers within 7 days prior to initiation of study treatment;

22. Vaccinated with live, attenuated vaccines within 6 months of enrollment;

23. Known or suspected allergies, hypersensitivity, or intolerance to azacitidine, golcadomide or its excipients;

24. Any known malabsorption syndrome or disease associated with malabsorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Modified Progression-Free Survival | From enrollment to end of follow-up period of Origina-ly-T (= maximum 2 years after enrollment)
  mPFS
Maximum Tolerated Dose | From enrollment to end of treatment of sub-study GolcAza (= maximum 2 years from enrollment)
  MTD
Recommended Phase II Dose | From enrollment to end of treatment of sub-study GolcAza (= maximum 2 years from enrollment)
  RP2D

CONTACTS AND LOCATIONS:
Overall Officials: François LEMONNIER, Pr, Principal Investigator — Hôpital Henri Mondor - Lymphoid Malignancies Unit
Locations (20):
- France (20):
  - Institut d'Hématologie de Basse Normandie - Service Hématologie (CHU Hôpital Côte de Nacre), Caen
  - CHU Estaing - Service Thérapie Cellulaire et Hématologie Clinique, Clermont-Ferrand
  - Hôpital Henri Mondor - Unité Hémopathies Lymphoïdes, Créteil
  - CHU Dijon Bourgogne - Service Hématologie Clinique, Dijon
  - CHU de Grenoble - Service Hématologie, La Tronche
  - CH du Mans - Centre de Cancérologie de la Sarthe - Service Hématologie, Le Mans
  - CHU de Lille - Hôpital Claude Huriez - Service des Maladies du Sang, Lille
  - Institut Paoli Calmettes - Service Hématologie, Marseille
  - CHU de Montpellier - Département d'Hématologie Clinique, Montpellier
  - CHU de Nantes - Service Hématologie, Nantes
  - Hôpital Necker - Service Hématologie Adultes, Paris
  - CHU de Bordeaux - Hôpital Haut-Lévêque - Centre François Magendie - Service d'Hématologie et Thérapie Cellulaire, Pessac
  - CHU Lyon-Sud - Hématologie Clinique, Pierre-Bénite
  - CHU de Poitiers - Hôpital de la Milétrie - Service d'Oncologie Hématologique et Thérapie Cellulaire, Poitiers
  - CHU Pontchaillou - Hématologie Clinique, Rennes
  - Centre Henri Becquerel - Service Hématologie, Rouen
  - Institut de Cancérologie et d'Hématologie Universitaire de Saint-Étienne - Service Hématologie, Saint-Etienne
  - CH de la Côte Basque - Service Hématologie, Saint-Jean-de-Luz
  - Institut de Cancérologie Strasbourg Europe - Service Hématologie, Strasbourg
  - CHRU Nancy - Hôpital Brabois - Service Hématologie, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No